CLINICAL TRIAL: NCT05301608
Title: Effects of Psilocybin on Electrophysiology and the Dynamic Content of Thought
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: IRB00251021
Record Dates: First submitted 2022-03-18; First posted 2022-03-29 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Healthy
Keywords: psilocybin; electroencephalography (EEG); magnetic resonance imaging (MRI); creativity; cognition
MeSH Terms: interventions — Psilocybin

STUDY DESIGN:
Intervention Model Description: All participants will receive all interventions, in counter-balanced order.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind, placebo-controlled, full cross-over masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Psilocybin First (Experimental): Psilocybin (10mg) will be administered one time orally as a capsule taken with water. Expected duration of acute effects is approximately 6 hours. After a period of a washout, participants will switch to the placebo intervention.
  Interventions: Drug: Psilocybin; Drug: Placebo
- Placebo First (Placebo Comparator): Participants will be administered placebo in a clinical setting. Placebo is administered orally as a capsule taken with water. After a period of a washout, participants will switch to the Psilocybin intervention.
  Interventions: Drug: Psilocybin; Drug: Placebo

INTERVENTIONS:
Drug: Psilocybin — The psilocybin used in this study is synthetically manufactured and formulated under current good manufacturing practices (cGMP). The active drug is encapsulated using a size 0 blue gelatin capsule and contains 10 mg of psilocybin.
  Other Names: 4-phosphoryloxy-N,N-dimethyltryptamine
Drug: Placebo — The placebo used in this study is microcrystalline cellulose, an inert substance, encapsulated using a size 0 blue gelatin capsule.

SUMMARY:
This research study will use computerized tasks, electroencephalography (EEG), and magnetic resonance imaging (MRI) to look at how the drug psilocybin, a naturally occurring compound contained in hundreds of species of psychoactive mushrooms, changes thoughts and brain activity.

DETAILED DESCRIPTION:
In this double-blind, placebo-controlled, within-subject, full cross-over study in healthy volunteers, computerized, electroencephalography (EEG), and magnetic resonance imaging (MRI) measures will be assessed to test the acute effects of a moderate dose of psilocybin (10 mg/70 kg) on creativity, the contents and dynamics of thought, memory, and shared vs individual brain response while viewing naturalistic stimuli. Understanding the acute psychological and neural effects of psychedelic drugs such as psilocybin may allow for future optimization of psychedelic medicine, as well as a deeper and more refined understanding of consciousness itself.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 75 years old
* Have given written informed consent
* Have at least a high-school level of education or equivalent (e.g. GED) and be fluent in English
* Be healthy and psychologically stable as determined by screening for medical and psychiatric problems via a personal interview, a medical questionnaire, a physical examination, an electrocardiogram (ECG), and routine medical blood and urinalysis laboratory tests
* Agree to consume approximately the same amount of caffeine-containing beverage (e.g. coffee, tea) that he/she consumes on a usual morning, before arriving at the research unit on the morning of the drug session day. If the participant does not routinely consume caffeinated beverages, he/she must agree not to do so on the session day.
* Agree to refrain from using any psychoactive drugs, including alcoholic beverages and nicotine, within 24 hours of each drug administration. The exception is caffeine.
* Agree not to take any "as-needed" medications on the mornings of drug sessions
* Agree not to take sildenafil (Viagra®), tadalafil, or similar medications within 72 hours of each drug administration.
* Agree that for one week before each drug session, he/she will refrain from taking any nonprescription medication, nutritional supplement, or herbal supplement except when approved by the study investigators. Exceptions will be evaluated by the study investigators and will include acetaminophen, non-steroidal anti-inflammatory drugs, and common doses of vitamins and minerals.
* Have used a psychedelic drug (e.g. lysergic acid diethylamide(LSD)/acid, psilocybin mushrooms, ayahuasca) at least five times in their lifetime.
* Proof of COVID-19 vaccination

Exclusion Criteria:

* Women who are pregnant (as indicated by a positive urine pregnancy test assessed at intake and before each drug session) or nursing; women who are of child-bearing potential and sexually active who are not practicing an effective means of birth control.
* Cardiovascular conditions: coronary artery disease, stroke, angina, uncontrolled hypertension, a clinically significant ECG abnormality (e.g. atrial fibrilation), artificial heart valve, or heart attack in the past year
* Epilepsy with history of seizures
* Insulin-dependent diabetes; if taking oral hypoglycemic agent, then no history of hypoglycemia
* Currently taking psychoactive prescription medication on a regular (e.g. daily) basis
* Currently taking on a regular (e.g. daily) basis any medications having a primary centrally-acting serotonergic effect, including mono-amine oxidase inhibitors (MAOIs). For individuals who have intermittent or "as needed" use of such medications, psilocybin sessions will not be conducted until at least five half-lives of the agent have elapsed after the last dose.
* More than 20% outside the upper or lower range of ideal body weight according to Metropolitan Life height and weight table
* Current or past history of meeting Diagnostic and Statistical Manual, version 5 (DSM-5) criteria for schizophrenia spectrum or other psychotic disorders (except substance/medication-induced or due to another medical condition)
* Current or past history within the last five years of meeting DSM-5 criteria for a moderate or severe alcohol or drug use disorder (excluding caffeine and nicotine)
* Have a first or second-degree relative with bipolar I disorder, schizophrenia spectrum, or other psychotic disorders (except substance/medication-induced or due to another medical condition)
* Has a psychiatric condition judged to be incompatible with establishment of rapport or safe exposure to psilocybin
* Has history of migraine, tension, or other recurring headaches.
* Head trauma, traumatic brain injury, or concussion with loss of consciousness for >2 minutes
* Contraindications for magnetic resonance imaging (MRI) (e.g. claustrophobia incompatible with MRI scanning, medical device or implant incompatible with MRI, prior history as a metal worker and/or certain metallic objects in the body)
* Left-handedness (assessed by the Edinburgh Handedness Inventory)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-03-03 (Actual); Primary Completion 2026-02-09 (Estimated); Study Completion 2026-06-09 (Estimated)

PRIMARY OUTCOMES:
Difference between drug conditions in the frequency of word use during free association tasks | 8 weeks
  Volunteers are instructed to either describe their interpretation of visual stimuli, verbalize a set of freely associated words, or reflect upon and describe out loud the thoughts that are occurring after presentation of short excerpts of popular music. Audio recordings of verbal responses from volunteers will be recorded, transcribed, and then submitted to automated text analysis and natural language processing analysis to compare the semantic content of responses between those that were provided during placebo and those that were provided during psilocybin conditions. The frequency of words that fall into a series of semantic categories (e.g. pronouns, adjectives, positive vs negative valence words) will be compared between drug conditions.
Sensitivity in distinguishing old versus newly presented visual stimuli | 8 weeks
  During drug administration sessions, volunteers will view a series of visual stimuli (words and images) and will be asked to read and remember each visual stimulus. The next day, volunteers will be presented with stimuli that were as well as stimuli that were not presented the previous day, and they will be asked to indicate the confidence with which they remember seeing the given stimulus before ("old") or not ("new"). Sensitivity in distinguishing between old and new words (d') will be calculated from receiver operator characteristic curve analysis of confidence ratings of "new" vs "old" judgements, and compared between drug conditions.
Accuracy in the remote associates task as assessed by total correct number of trials | 8-week study period
  Participants will be presented with three words that are only remotely related to each other (e.g., falling, actor, dust) and ask them to generate a fourth word (e.g., star) that relates to all three words. Total correct number of trials will be compared between drug conditions.
Accuracy in the alternative uses task | 8-week study period
  The Alternative Uses Task assesses the extent one can generate novel uses for presented stimuli (e.g. a brick, or a paper clip). The total number of responses and the number of uniquely novel uses that were generated will be compared between drug conditions.
Alpha band power in EEG record | 8-week study period
  Continuous EEG recordings will be analyzed using spectral decomposition, and the time course of average power in the alpha frequency band will be compared between drug conditions.
Reliability of whole-brain response while watching videos | 8-week study period
  Volunteers will be presented with videos during scanning in the second two drug administration sessions. These will be otherwise unremarkable 6-15 minute videos of natural scenes, human interactions, or narrative stories. We will calculate correlations in measured brain response across subjects, moment-by-moment, which yields a measure of reliability of response to these videos across the brain. This reliability map will be compared between drug conditions.

CONTACTS AND LOCATIONS:
Overall Officials: Frederick S Barrett, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Center for Psychedelic and Consciousness Research, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual participant data will be made available in public databases (e.g. OSF).
Supporting Information: Study Protocol, ICF, Analytic Code
Time Frame: Data will be made available in public databases after study findings have been published.
Access Criteria: Data will be accessible to qualified researchers.